CLINICAL TRIAL: NCT03780855
Title: Preliminary Evaluation of the Safety and Effectiveness of the Bionic Nerve Scaffold With Longitudinally Oriented Microchannels in Clinical Application
Brief Title: Preliminary Evaluation of the Clinical Safety and Effectiveness of the Bionic Nerve Scaffold
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Xijing Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: KY20172005-1
Record Dates: First submitted 2018-11-26; First posted 2018-12-19 (Actual); Last update posted 2018-12-19 (Actual); Status verified 2017-12

CONDITIONS: Peripheral Nerve Injuries
Keywords: scaffold; Peripheral nerve injures; repair; safety; effectiveness
MeSH Terms: conditions — Peripheral Nerve Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- nerve scaffold group (Experimental): the experimental group of cases with peripheral sensory nerve injuries will be treated with nerve scaffold.
  Interventions: Device: nerve scaffold
- non-nerve scaffold group (No Intervention): the control group of cases will be treated without nerve scaffold.

INTERVENTIONS:
Device: nerve scaffold — It is a new kind of nerve scaffold with the microstructure of longitudinally oriented microchannels. It's made of collagen as the main raw material.
  Arms: nerve scaffold group

SUMMARY:
The objective of the study is to preliminarily evaluate the clinical safety and effectiveness of the bionic nerve scaffold with longitudinally oriented microchannels. 10 patients with peripheral sensory nerve defects will be involved and divided into 2 groups: the experimental group is treated with the nerve scaffold, and the control group without that. Then follow the cases up and draw conclusion according to the results of observation and examination.

DETAILED DESCRIPTION:
The objective of the study is to preliminarily evaluate the clinical safety and effectiveness of the bionic nerve scaffold with longitudinally oriented microchannels developed in the Department of Orthopaedics in Xijing hospital in repairing the peripheral nerve defect. According to the inclusion and exclusion criteria, 10 patients with peripheral sensory nerve defects of 1 to 3 cm in size will be involved. Divided them into 2 groups. The experimental group of 5 cases will be treated with the nerve scaffold, and the control group without that. Then follow the cases up at about 2 weeks, 3 months and 6 months after surgery. Observe the condition of the healing of the local wound and the whole body of the 10 patients. Examine the blood routine and biochemical indexes of the experimental group. Sensory recovery of injured nerves will be tested at about 3 months and 6 months after surgery. Record the results in the case report forms. Analyze the data statistically and draw conclusion.

ELIGIBILITY:
Inclusion Criteria:

* age from 18-50 yeas old, male or female, course of disease is within one year;
* good heart, liver and kidney function;
* with peripheral sensory nerve defects of 1-3 cm in size, and willing to repair it with the nerve scaffold;
* no significant damage existing in the skin and soft tissue in the operative region
* have signed the informed consent form
* good adherence and willing to return for follow-up visits as required.

Exclusion Criteria:

* with acute or severe infection
* suffering from serious primary diseases of heart, brain, liver and kidney, blood system, endocrine system and so on, and can not tolerate surgery
* with histories of peripheral vascular disease, immunological disorder chronic alcoholism, and drug abuse and so on
* with family history of genetic
* allergic to collagen and chitosan
* pregnancy and lactating women
* serious damage existing in the skin and soft tissue in the operative region
* bad adherence and can not return for follow-up visits on time as required

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 10 (Estimated)
Dates: Start 2017-06-14 (Actual); Primary Completion 2019-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Observing the condition of the healing of local wound with the naked eye at 2 weeks after operation，including redness, exudation and ulceration. | 2 weeks after operation
  The condition of the healing of local wound will be observed by the designated doctor with the naked eye to see if there is redness, exudation or ulceration. And then the condition will be recorded.
Learning about patients' systemic reactions by asking them at 2 weeks after operation, including fever, nausea, vomiting and skin itching. | 2 weeks after operation
  The patients will be asked if there is systemic discomfort or any other bad reactions during the 2 weeks, including fever, nausea, vomiting and skin itching. And then the condition will be recorded.
Test of white blood cell count at 2 weeks after operation | 2 weeks after operation
  Blood routine test will be conducted in our hospital. And then the value of white blood cell count will be recorded.
Test of lymphocyte count at 2 weeks after operation | 2 weeks after operation
  Blood routine test will be conducted in our hospital. And then the value of lymphocyte count will be recorded.
Test of red blood cell count at 2 weeks after operation | 2 weeks after operation
  Blood routine test will be conducted in our hospital. And then the value of red blood cell count will be recorded.
Test of hemoglobin concentration at 2 weeks after operation | 2 weeks after operation
  Blood routine test will be conducted in our hospital. And then the value of hemoglobin concentration will be recorded.
Test of platelet count at 2 weeks after operation | 2 weeks after operation
  Blood routine test will be conducted in our hospital. And then the value of platelet count will be recorded.
Test of alanine aminotransferase at 2 weeks after operation | 2 weeks after operation
  Liver function test will be conducted in our hospital. And then the value of alanine aminotransferase will be recorded.
Test of aspartate aminotransferase at 2 weeks after operation | 2 weeks after operation
  Liver function test will be conducted in our hospital. And then the value of aspartate aminotransferase will be recorded.
Test of serum creatinine at 2 weeks after operation | 2 weeks after operation
  Kidney function test will be conducted in our hospital. And then the value of serum creatinine will be recorded.
Test of blood urea nitrogen at 2 weeks after operation | 2 weeks after operation
  Kidney function test will be conducted in our hospital. And then the value of blood urea nitrogen will be recorded.
Test of prothrombin time at 2 weeks after operation | 2 weeks after operation
  Hemagglutination series test will be conducted in our hospital. And then the value of prothrombin time will be recorded.
Test of activated partial thromboplastin time at 2 weeks after operation | 2 weeks after operation
  Hemagglutination series test will be conducted in our hospital. And then the value of activated partial thromboplastin time will be recorded.
Test of thrombin time at 2 weeks after operation | 2 weeks after operation
  Hemagglutination series test will be conducted in our hospital. And then the value of thrombin time will be recorded.
Examination of the position sense at 3 months after operation | 3 months after operation
  The position sense of the area innervated by the repaired nerve will be examined by the designated doctor, which is a kind of deep sense.
Examination of the movement sense at 3 months after operation | 3 months after operation
  The movement sense of the area innervated by the repaired nerve will be examined by the designated doctor, which is another kind of deep sense.
Examination of the sense of light touch at 3 months after operation | 3 months after operation
  The sense of light touch of the area innervated by the repaired nerve will be examined by the designated doctor, which is one of the superficial sense categories.
Examination of the sense of pain at 3 months after operation | 3 months after operation
  The sense of pain of the area innervated by the repaired nerve will be examined by the designated doctor, which is another one of the superficial sense categories.
Examination of the sense of temperature at 3 months after operation | 3 months after operation
  The sense of temperature of the area innervated by the repaired nerve will be examined by the designated doctor, which also belongs to the superficial sense categories.
Examination of static two-point discrimination at 3 months after operation | 3 months after operation
  The static two-point discrimination of the area innervated by the repaired nerve will be examined by the designated doctor.
Test of white blood cell count at 3 months after operation | 3 months after operation
  Blood routine test will be conducted in our hospital. And then the value of white blood cell count will be recorded.
Test of lymphocyte count at 3 months after operation | 3 months after operation
  Blood routine test will be conducted in our hospital. And then the value of lymphocyte count will be recorded.
Test of red blood cell count at 3 months after operation | 3 months after operation
  Blood routine test will be conducted in our hospital. And then the value of red blood cell count will be recorded.
Test of hemoglobin concentration at 3 months after operation | 3 months after operation
  Blood routine test will be conducted in our hospital. And then the value of hemoglobin concentration will be recorded.
Test of platelet count at 3 months after operation | 3 months after operation
  Blood routine test will be conducted in our hospital. And then the value of platelet count will be recorded.
Test of alanine aminotransferase at 3 months after operation | 3 months after operation
  Liver function test will be conducted in our hospital. And then the value of alanine aminotransferase will be recorded.
Test of aspartate aminotransferase at 3 months after operation | 3 months after operation
  Liver function test will be conducted in our hospital. And then the value of aspartate aminotransferase will be recorded.
Test of serum creatinine at 3 months after operation | 3 months after operation
  Kidney function test will be conducted in our hospital. And then the value of serum creatinine will be recorded.
Test of blood urea nitrogen at 3 months after operation | 3 months after operation
  Kidney function test will be conducted in our hospital. And then the value of blood urea nitrogen will be recorded.
Test of prothrombin time at 3 months after operation | 3 months after operation
  Hemagglutination series test will be conducted in our hospital. And then the value of prothrombin time will be recorded.
Test of activated partial thromboplastin time at 3 months after operation | 3 months after operation
  Hemagglutination series test will be conducted in our hospital. And then the value of activated partial thromboplastin time will be recorded.
Test of thrombin time at 3 months after operation | 3 months after operation
  Hemagglutination series test will be conducted in our hospital. And then the value of thrombin time will be recorded.
Examination of the position sense at 6 months after operation | 6 months after operation
  The position sense of the area innervated by the repaired nerve will be examined by the designated doctor, which is a kind of deep sense.
Examination of the movement sense at 6 months after operation | 6 months after operation
  The movement sense of the area innervated by the repaired nerve will be examined by the designated doctor, which is another kind of deep sense.
Examination of the sense of light touch at 6 months after operation | 6 months after operation
  The sense of light touch of the area innervated by the repaired nerve will be examined by the designated doctor, which is one of the superficial sense categories.
Examination of the sense of pain at 6 months after operation | 6 months after operation
  The sense of pain of the area innervated by the repaired nerve will be examined by the designated doctor, which is another one of the superficial sense categories.
Examination of the sense of temperature at 6 months after operation | 6 months after operation
  The sense of temperature of the area innervated by the repaired nerve will be examined by the designated doctor, which also belongs to the superficial sense categories.
Examination of static two-point discrimination at 6 months after operation | 6 months after operation
  The static two-point discrimination of the area innervated by the repaired nerve will be examined by the designated doctor.
Test of white blood cell count at 6 months after operation | 6 months after operation
  Blood routine test will be conducted in our hospital. And then the value of white blood cell count will be recorded.
Test of lymphocyte count at 6 months after operation | 6 months after operation
  Blood routine test will be conducted in our hospital. And then the value of lymphocyte count will be recorded.
Test of red blood cell count at 6 months after operation | 6 months after operation
  Blood routine test will be conducted in our hospital. And then the value of red blood cell count will be recorded.
Test of hemoglobin concentration at 6 months after operation | 6 months after operation
  Blood routine test will be conducted in our hospital. And then the value of hemoglobin concentration will be recorded.
Test of platelet count at 6 months after operation | 6 months after operation
  Blood routine test will be conducted in our hospital. And then the value of platelet count will be recorded.
Test of alanine aminotransferase at 6 months after operation | 6 months after operation
  Liver function test will be conducted in our hospital. And then the value of alanine aminotransferase will be recorded.
Test of aspartate aminotransferase at 6 months after operation | 6 months after operation
  Liver function test will be conducted in our hospital. And then the value of aspartate aminotransferase will be recorded.
Test of serum creatinine at 6 months after operation | 6 months after operation
  Kidney function test will be conducted in our hospital. And then the value of serum creatinine will be recorded.
Test of blood urea nitrogen at 6 months after operation | 6 months after operation
  Kidney function test will be conducted in our hospital. And then the value of blood urea nitrogen will be recorded.
Test of prothrombin time at 6 months after operation | 6 months after operation
  Hemagglutination series test will be conducted in our hospital. And then the value of prothrombin time will be recorded.
Test of activated partial thromboplastin time at 6 months after operation | 6 months after operation
  Hemagglutination series test will be conducted in our hospital. And then the value of activated partial thromboplastin time will be recorded.
Test of thrombin time at 6 months after operation | 6 months after operation
  Hemagglutination series test will be conducted in our hospital. And then the value of thrombin time will be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Zhuo j Luo, MD, Study Chair — Xijing Hospital; Rui Cong, MD, Study Director — Xijing Hospital
Locations (1):
- Xijing Hospital, Xi'an, Shaanxi, China